CLINICAL TRIAL: NCT04795583
Title: A Randomized Clinical Trial Comparing 7 Days Treatment With Corticosteroids Versus Placebo for Early COVID-19
Brief Title: Corticosteroids for COVID-19
Acronym: CORE-COVID
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Funding Issues
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00001
Record Dates: First submitted 2021-03-10; First posted 2021-03-12 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2021-06

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Prednisone (Experimental): Treatment adjusted by weight. Prednisone 25 mg capsules:
  * ≤ 50kg = 2 capsules QD x 7 days (maximum dose = 50mg/day)
  * 50 - 80kg = 3 capsules QD x 7 days (maximum dose = 75mg/day)
  * > 80kg = 4 capsules QD x 7 days (maximum dose = 100mg/day)
  Interventions: Drug: Prednisone; Device: Point of Care testing device for C-reactive protein
- Placebo (Placebo Comparator): Capsules with the same appearance as Prednisone
  Interventions: Device: Point of Care testing device for C-reactive protein

INTERVENTIONS:
Drug: Prednisone — Prednisone 25 mg capsules
  Arms: Prednisone
Device: Point of Care testing device for C-reactive protein — Determination of C-reactive protein blood levels by point of care testing device

SUMMARY:
This trial is an interventional, randomized, placebo-controlled, adaptive clinical trial in outpatients with symptomatic microbiologically-confirmed SARS-CoV-2, in stable clinical condition, and increased levels of serum C-reactive protein. The hypothesis of this study is that early administration of prednisone for 7 days in patients with evidence of increased C-reactive protein will decrease the progression of COVID-19, prevent clinical deterioration, and hospital admission. Objectives: Primary Objective: To evaluate if early administration of corticosteroids in non-hospitalized participants with proven SARS-CoV-2 infection with compatible clinical symptoms and increased C-reactive protein can prevent hospital admission or early death

DETAILED DESCRIPTION:
The proposed trial is an interventional, randomized, placebo-controlled, adaptive clinical trial in outpatients with symptomatic microbiologically-confirmed SARS-CoV-2, in stable clinical condition, and increased levels of serum C-reactive protein.

Potential participants will be identified via Public Health after a diagnosis of SARS-CoV-2 infection is made either by positive nucleic acid testing or by antigen detection, from a nasal or pharyngeal swab. These study candidates will be asked for permission to be contacted. If this person agrees, a research collaborator will contact the potential participant by phone call. During this phone call, verbal informed consent to be included in the study will be requested.

After inclusion in the study, participants will be divided into two groups with the below follow-up outline:

* Group 1 non-RCT: Asymptomatic participants (no symptoms of early COVID-19). These participants will be followed by phone call every 48 hours for 14 days. If asymptomatic participants develop clinical symptoms of early COVID-19 during follow-up (pre-symptomatic COVID-19), they will be transferred to Group 2. Otherwise, study for this group will end at the 14 days timepoint with the exception 20 participants who consent to partake in the pulmonary evaluation at 12 weeks (tertiary/exploratory objective, see sections 3.1 and 7.1).
* Group 2 non-RCT: Participants with symptoms of early COVID-19 will undergo full follow-up every 48 hours for 4 visits (8 days) which will consist of:

  * Review of clinical symptoms by phone call.
  * Oxygen saturation.
  * C-reactive protein in blood.

The strategy for the follow-up visits is described below. Participants in this group who present with the inclusion criteria and without exclusion criteria (section 1.5) will be asked to join the randomized control trial. Otherwise, study for this group will end at the 8 days time point with the exception of 20 participants who consent to partake in the pulmonary evaluation at 12 weeks (tertiary/exploratory objective, see sections 3.1 and 7.1).

Study visits:

Monitoring of C-reactive protein and oxygen saturation will be evaluated at the participant's home following a COVID-19 safe procedure. C-reactive protein will be determined by a point-of-care diagnostic device (Afinion[TM] 2 Analyzer, Abbott Laboratories, USA; Health Canada Regitration number 99614) using C-reactive protein cartridges and controls by the same manufacturer (Afinion CRP and Afinion CRP control Health Canada Registration number 98995). More information of the point-of-care device can be found at: https://www.globalpointofcare.abbott/en/product-details/afinion2-analyzer.html). A kit with all the necessary materials (gloves, lancet, alcohol scrubs, pulse oximeter (ToronTek-E400, Health Canada Registration number: 90629) and AfinionTM C-reactive protein cartridges) will be placed at the front door of the participant's home. In the case of long-term care facilities, nursing homes or other facilities with healthcare workers, the kit will be provided to the participant's main caregiver. The research associate (research coordinator, research assistant or medical student) will never be in contact with the participant or relatives and will always wear a mask and gloves to manipulate the material.

An educational video will be offered to participants to self-perform blood drop collection to the integrated capillary system. Those patients unable to perform self-collection of blood drop will be offered to remain in the study to know the evolution of clinical symptoms and outcome.

In each visit, a kit will be delivered to the participant's home by a research coordinator or research assistant. The content of the kit for each visit will contain the following items.

1. Pulse oximeter.
2. Surgical mask.
3. Alcohol pads (x2).
4. Single-use lancet (Unistik 3, Owen Mumford Ltd, Health Canada Licence No.: 9790) (x2).
5. Afinion 2 CRP cartridge.
6. Paper sheet.
7. Pen.

In the first visit, the kit will contain a 50 mL bottle of hand sanitizer and a 1-liter sharp container that the participant will retain for the following visits. Briefly, the patient will be instructed to wash her/his hands before collecting the kit. Before touching any other item, the participant will put on the surgical mask. The next step will be to register the oxygen saturation using the pulse oximeter and will register the value on the paper sheet. After cleaning the tip of a finger with an alcohol pad, the participant will obtain a blood drop and load the capillary of the C-reactive cartridge. After completing this task, the visit will be completed and the participant will return the kit containing the pen, paper sheet, Afinion 2 CRP cartridge and pulse oximeter. The participant will be instructed to deposit the used lancet in the sharp container.

Intervention: Eligible participants who sign informed consent for the RCT will be randomized at a ratio of 1:1 to:

* Oral prednisone in 25mg capsules with a dosage determined according to weight range for 7 days.
* Oral placebo capsules with the same appearance daily for 7 days.

Follow-up of RCT participants post-randomization and end of study (Figure 1, Table 2):

1. During intervention (Day 0 to 7 post-randomization):

   i. A baseline questionnaire (EQ-5D-5L) for state of patient health will be collected at day 0.

   ii. Clinical monitoring by phone call at day 3 and end of treatment (day 7). iii. C-reactive protein levels and oxygen saturation at the end of treatment (day 7) collected as described above.
2. After intervention (Week 1 to 12 post-randomization):

   i. Once treatment is completed, follow up will be performed by phone calls on a weekly basis until week 12 post-randomization (end of study).
3. End of study (Week 12 post-randomization). Visit at the post-COVID clinic. i. Participants will be asked to complete the EQ-5D-5L questionnaire and the Post-COVID Functional Status (PCFS) scale.

ii. Spirometry: FEV1, FVC, FEV1/FVC. iii. 6-minute walking test.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Microbiologically-confirmed SARS-CoV-2.
3. Clinical symptoms compatible with COVID-19 for 14 days or less before randomization.
4. Oxygen saturation ≥ 95%.
5. Protein C-reactive in blood performed by point-of-care testing ≥ 20 mg/L.
6. Signed informed consent.

Exclusion Criteria:

1. Oxygen requirement at home due to chronic lung disease.
2. Patients with immunosuppression or immunosuppressive therapies defined as:

   * Cancer on active chemotherapy.
   * Stem cell transplant in the previous 6 months.
   * Neutrophil count < 1000 cells/mm3.
   * Chronic treatment with immunosuppressive therapy, except for low-dose (≤10 mg daily) prednisone or equivalent dose of other corticosteroids.
   * HIV-infected patients with CD4 < 200 x 106/L.
   * Diagnosis with primary immunodeficiencies.
3. Chronic liver damage Child-Pugh C.
4. Chronic underlying process with suspected life expectancy less than 12 weeks.
5. Uncontrolled diabetes mellitus at screening, defined as no blood glucose testing or any blood glucose level higher than 14 mmol/L (or 250 mg/dL) in the last 14 days.
6. Diagnosis of any form of psychosis without receiving appropriate treatment.
7. Pregnancy at time of randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Hospital admission or death in the first 2 weeks after randomization | 14 days
  Need to be admitted to hospital or death during the first 2 weeks after randomization

SECONDARY OUTCOMES:
Hospitalization at 30 days | 30 days
  Need of hospital admission in the first 30 days after randomization
Mortality at 30 days | 30 days
  Death in the first 30 days after randomization
Serious adverse events at 30 days | 30 days
  Occurrence of SAEs in the first 30 days after randomization
Death at week 12 | Week 12
  Death in the first 12 weeks after randomization
Duration of symptoms | Week 12
  COVID-19 symptoms duration in days

OTHER OUTCOMES:
Long COVID-19 | 12 weeks
  Persistent symptoms of COVID-19 at week 12 of randomization

CONTACTS AND LOCATIONS:
Locations (2):
- Clinica de la Mujer, Bogotá, Colombia
- ABC Medical Center, Mexico City, Mexico